CLINICAL TRIAL: NCT04868136
Title: The Effects of a Dynamic Warm up on the Immune Response to Exercise in Lower Fit and Higher Fit Adults
Brief Title: Effects of a Warm-up on Immune Response to Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Emily C Lavoy, Assistant Profesor, University of Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00000990
Record Dates: First submitted 2021-04-25; First posted 2021-04-30 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Physiological and Psychological Responses to Exercise
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized cross-over study with two conditions. Randomization was stratified by sex
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm-up, then no warm-up (Experimental): Participants' visit 2 included 10 minutes of gradually increasing intensity prior to the 30 minute exercise session. Participants' visit 3 consisted of the 30 minute exercise session without a warm-up.
  Interventions: Behavioral: Exercise
- No warm-up, then warm-up (Experimental): Participants' visit 2 consisted of the 30 minute exercise session without a warm-up. Participants' visit 3 included 10 minutes of gradually increasing intensity prior to the 30 minute exercise session.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — 30 minutes of exercise at 80% of maximum predicted heart rate performed on an indoor stationary bicycle. Exercise was preceded by 10 min of gradually increasing cycling intensity in one of two exercise trials
  Other Names: Cardiorespiratory exercise

SUMMARY:
This randomized cross-over study compares two identical cardiorespiratory exercise bouts, differing only in the inclusion or exclusion of a dynamic period of increasing exercise intensity prior to the exercise bout. Planned comparisons include physiological responses and perceived effort during exercise, leukocyte mobilization, and mood between the two exercise sessions.

DETAILED DESCRIPTION:
Physically active adult men and women are asked to complete three study visits to the laboratory. On Visit 1, participants provide informed consent and are screened for study inclusion criteria: being between 18 and 40 years of age, a non-smoker, not pregnant, free of disease impacting exercise performance or immunity, and performing at least one hour per week of vigorous exercise training (any modality) for at least the prior six months. Participants also complete an incremental submaximal exercise test on a stationary bicycle. The results of this test are used to calculate the resistance corresponding to 80% of estimated maximal heart rate. Participants return within 2-14 days for Visits 2 and 3. These visits consist of 30 min of bicycling at this resistance. One visit included a 10 min dynamic warm-up prior to the exercise bout. Participants were stratified by sex and randomized such that half of the men and women completed the exercise trial with warm-up during Visit 2.

Heart rate, perceived exertion, and wattage are recorded during each minute of the exercise bouts. Participants donate blood before, immediately after, and 1h after each exercise. Blood is analyzed by flow cytometry to characterize leukocyte subsets. After each exercise session, participants complete surveys assessing mood and affect.

Physiological, immunological, and psychological parameters recorded will be compared within participants between the two experimental exercise sessions using appropriate statistical tests. p<0.05 will be accepted as significant.

ELIGIBILITY:
Inclusion Criteria:

* identifies as exercising 1-3 hours per week or more than 6 hours per week, on average (last 6 months)
* meets American College of Sports Medicine criteria for participation in exercise

Exclusion Criteria:

* underlying medical problems that contraindicate supervised high intensity exercise
* past or present history of autoimmune disease, HIV, hepatitis, stroke, or cardiovascular disease
* chronic/debilitating arthritis
* central or peripheral nervous disorders
* asthma, emphysema, or bronchitis
* bedridden in the past three months
* history of blood clotting disorders
* administration of any medication that might affect physiological response to exercise
* functional or cognitive impairment that would limit exercise performance or prohibit informed consent
* having any common-cold or influenza like symptoms (scratchy throat, runny nose, inflamed sinuses, frequent sneezing or coughing) in the last 2 weeks
* pregnancy
* tobacco use

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Heart rate during exercise | Minutes 1-30 of exercise, recordings made each minute
  Heart rate in beats per minute
Perceived exertion during exercise | Minutes 1-30 of exercise, recordings made each minute
  Rating of perceived exertion measured using the Borg 6-20 scale
Power during exercise | Minutes 1-30 of exercise, recordings made each minute
  Wattage produced on stationary bicycle
Monocyte mobilization by exercise | Change from resting levels of monocytes after exercise
  Number of peripheral blood monocytes
Natural Killer cell mobilization by exercise | Change from resting levels of natural killer cells after exercise
  Number of peripheral blood natural killer cells
CD4 T cell mobilization by exercise | Change from resting levels of CD4 T cells after exercise
  Number of peripheral blood CD4 T cells
CD8 T cell mobilization by exercise | Change from resting levels of CD8 T cells after exercise
  Number of peripheral blood CD8 T cells

SECONDARY OUTCOMES:
Mood after exercise | Measured within 10 minute of end of exercise session
  Mood dimensions characterized by Profile of Mood Survey
Affect after exercise | Measured within 10 minute of end of exercise session
  Affect characterized by Positive and Negative Affect Schedule

CONTACTS AND LOCATIONS:
Overall Officials: Emily C LaVoy, PhD, Principal Investigator — University of Houston
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data that underlie results in a publication will be made available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Will be available upon publication
Access Criteria: Requests should be sent to and will be reviewed by the principle investigator